CLINICAL TRIAL: NCT03064191
Title: Influence of Calcium Hydroxide Chlorhexidine Combination vs. Calcium Hydroxide as an Intra Canal Medicaments on Postoperative Flare -up Following Two-Visits Endodontic Retreatment Cases: Single Blinded Randomized Clinical Trial
Brief Title: Influence of Intra Canal Medications on Postoperative Flare-up in Endodontic Re-treatment Cases
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: rayan rabie dahab (Other)
Collaborators: Cairo University (Other)
Responsible Party: Sponsor-Investigator, rayan rabie dahab, principal investigator, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEBD-CU-2017-02-11
Record Dates: First submitted 2017-02-16; First posted 2017-02-24 (Actual); Last update posted 2017-09-12 (Actual); Status verified 2017-09

CONDITIONS: Postoperative Pain; Pain, Dental
Keywords: intra-canal medications
MeSH Terms: conditions — Pain, Postoperative; Toothache | interventions — Calcium Hydroxide

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- calcium hydroxide chlorhexidine (Active Comparator): intervention: calcium hydroxide chlorhexidine combination an intra-canal medication composed of calcium hydroxide powder and chlorhexidine solution as a combination to be administered as intra-canal paste for decreasing postoperative symptoms
  Interventions: Combination Product: calcium hydroxide chlorhexidine combination
- calcium hydroxide (Active Comparator): intervention: calcium hydroxide an intra-canal medicament composed of calcium hydroxide paste for decreasing postoperative symptoms and signs .
  Interventions: Other: calcium hydroxide intra-canal medicament

INTERVENTIONS:
Combination Product: calcium hydroxide chlorhexidine combination — Endodontic intra-canal medicament used for decreasing postoperative signs ans symptoms
  Other Names: intra-canal medicament combination
  Arms: calcium hydroxide chlorhexidine
Other: calcium hydroxide intra-canal medicament — Endodontic intra-canal medicament used for decreasing postoperative signs and symptoms.
  Other Names: calcium hydroxide, gold standard intra-canal medicament
  Arms: calcium hydroxide

SUMMARY:
Is to evaluate the influence of the calcium hydroxide / chlorhexidine combination and calcium hydroxide alone as an intra-canal medication in postoperative flare-up in two visits endodontic retreatment cases

DETAILED DESCRIPTION:
Problem: patient needs retreatment Intervention: calcium hydroxide chlorhexidine combination as an intra-canal medicament Control: calcium hydroxide alone as an intra-canal medicament Outcome: postoperative flare-up (pain and swelling) Time: after 7 days from 1st visit. population will be examined:

1. Patients' needs retreatment.
2. Patients in good health with no systemic disease (American Society of Anesthesiologists Class II)
3. Age range is between 20 and 50 years.
4. Patients who can understand the categorical tool (points)for measurement
5. Patients able to sign informed consent.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients' needs retreatment.
* 2. Patients in good health with no systemic disease (American Society of Anesthesiologists Class II)
* 3. Age range is between 20 and 50 years.
* 4. Patients who can understand the categorical tool (points)for measurement
* 5. Patients able to sign informed consent.

Exclusion Criteria:

* 1) Complicating systemic disease
* 2) Having severe pain and/or acute apical abscesses
* 3) Being under 18 years of age
* 4) Using antibiotics or corticosteroids,
* 5) having multiple teeth that required retreatment to eliminate the possibility of pain referral
* 6) Having root canals that could not be treated well with initial root canal treatment.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2017-09 (Estimated); Primary Completion 2018-03-13 (Estimated); Study Completion 2018-04-13 (Estimated)

PRIMARY OUTCOMES:
measuring patients postoperative pain and swelling following endodontic re-treatment sessions using Categorical (4 points) unit using questionnaire. | 7 days between the 2 visits ( one week)
  postoperative pain and swelling will be measured by:Categorical (4 points). The incidence of postoperative discomfort was recorded and expressed as numbers and percentages
  Subjectively into 4 points:
  1. no pain
  2. Mild pain: recognizable but not discomforting pain that required no analgesics.
  3. Moderate pain: discomforting but bearable pain(analgesics if used were effective in relieving pain)
  4. Severe pain: difficult to bear (analgesics were effective in relieving pain). Patients with severe postoperative pain and/or occurrence of swelling were classified as flare-ups.3 Objectively : percussion test

CONTACTS AND LOCATIONS:
Locations (1):
- Univeristy of Cairo, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided